CLINICAL TRIAL: NCT00659789
Title: A Phase II, Randomized, Double-blind, Multicenter, Immunogenicity Study of Vacc-4x Versus Placebo in Patients Infected With HIV-1 Who Have Maintained an Adequate Response to ART
Brief Title: Immunogenicity Study of Vacc-4x Versus Placebo in Patients Infected With HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bionor Immuno AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-BI Vacc-4x 2007/1; 2007-006302-13 (EudraCT Number); 13619 (Other: FDA IND)
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Results first posted 2017-01-05 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-11

CONDITIONS: HIV I Infection
MeSH Terms: interventions — Vacc-4x

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vacc-4x (Experimental): Vacc-4x reconstituted in sterile water (0.1 mL) at a dose of 1.2mg per intradermal administration. Participants are given a total of 6 immunizations over 18 weeks (weeks 1, 2, 3, 4, 16, 18). Recombinant human granulocyte macrophage colony stimulating factor (rhuGM-CSF) Leukine (0.06mg in 0.1 mL) administered intradermally is used as a local adjuvant.
  Interventions: Drug: Vacc-4x
- Placebo (Placebo Comparator): Placebo injections consisting of sterile water (0.1 mL) in place of Vacc-4x. Placebo injections consisting of sterile water (0.1 mL) in place of Leukine.
  Interventions: Drug: Sterile water

INTERVENTIONS:
Drug: Vacc-4x — Vacc-4x is a peptide-based HIV immunotherapy administered intradermally. Vacc-4x peptides are reconstituted in sterile water.
  Other Names: Combination of Vacc-10, Vacc-11, Vacc-12 and Vacc-13.
  Arms: Vacc-4x
Drug: Sterile water — Sterile water is used in place of Vacc-4x and in place of Leukine
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Current management of HIV infection includes anti-retroviral therapy (ART). ART cannot cure the infection, making it a life-long treatment that requires sustained patient compliance and imposes significant individual and societal financial burdens on healthcare services. Furthermore, ART side effects often require medication that increases the inconveniences and financial burdens of HIV management. Of further concern is the emergence of viruses resistant to ART that can result in treatment failure.

ART-free periods could provide substantial benefit. Vacc-4x is a peptide-based HIV immunotherapy that is proposed for prolongation of ART-free periods. The purpose of this study is to determine whether Vacc-4x immunotherapy can give safe ART-free period.

DETAILED DESCRIPTION:
Current management of HIV infection includes anti-retroviral therapy (ART). ART cannot cure the infection, making it a life-long treatment that requires sustained patient compliance and imposes significant individual and societal financial burdens on healthcare services. Furthermore,ART side effects often require medication that increases the inconveniences and financial burdens of HIV management. Of further concern is the emergence of viruses resistant to ART that can result in treatment failure.

ART-free periods could provide substantial benefit. Vacc-4x is a peptide-based HIV immunotherapy that is proposed for prolongation of ART-free periods. The purpose of this study is to determine whether Vacc-4x immunotherapy can give safe ART-free period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55
* HIV positive at least one year
* Clinically stable on ART for at least six months
* Documented viral load less than 50 copies/mL for the last six months
* Documented prestudy CD4 cell count equal or more than 400x10exp6/L
* Nadir CD4 cell count equal or more than 200x10exp6/L
* Signed informed consent

Exclusion Criteria:

* Reported pre-study AIDS-defining illness within the previous year
* Malignant disease
* On chronic treatment with immuno-suppressive therapy
* Unacceptable values of hematology and clinical chemistry parameters
* Current chronic infection such as HCV and HBV or active tuberculosis
* Pregnant or breastfeeding women
* Not using safe contraceptive methods
* Participation in other clinical trial
* Incapability of compliance

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 137 (Actual)
Dates: Start 2008-08; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Pollard, MD, Principal Investigator — University of California at Davis, USA; Jürgen Rochstroh, MD, Principal Investigator — Universitätsklinikum Bonn, Germany
Locations (18):
- United States (5):
  - UCLA CARE Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - University of Miami School of Medicine, Miami, Florida
  - Northwestern University Division of Infectious Diseases, Chicago, Illinois
- Germany (6):
  - EPIMED GmbH, Berlin, State of Berlin
  - Charité Universitätsmedizin Berlin, Berlin, State of Berlin
  - Universitätsklinikum Bonn, Bonn
  - Klinik I für Innere Medizin Klinikum Der Universität zu Köln, Cologne
  - ifi - Studien und Projekte GmbH, an der Asklepios-Klinik St. George, Hamburg
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
- Istituto San Raffaele, Milan, Italy
- Spain (3):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Clinic i Provincial, Barcelona
  - Unidad de VIH, Hospital de Bellvitge, Calle Feixa Llarga s/n, Hospitalet de Llobregat., Barcelona
- United Kingdom (3):
  - Brighton and Sussex University Hospital, HIV/GUM Research, Elton John Centre, Brighton
  - Chelsea and Westminster Hospital, London
  - Harrison Wing St Thomas' Hospital, London

IPD SHARING:
Plan to Share IPD: No
Participants have not provided informed consent for their anonymized individual data to be made available beyond that described in the patient information sheet.

REFERENCES:
- [Derived] Pollard RB, Rockstroh JK, Pantaleo G, Asmuth DM, Peters B, Lazzarin A, Garcia F, Ellefsen K, Podzamczer D, van Lunzen J, Arasteh K, Schurmann D, Clotet B, Hardy WD, Mitsuyasu R, Moyle G, Plettenberg A, Fisher M, Fatkenheuer G, Fischl M, Taiwo B, Baksaas I, Jolliffe D, Persson S, Jelmert O, Hovden AO, Sommerfelt MA, Wendel-Hansen V, Sorensen B. Safety and efficacy of the peptide-based therapeutic vaccine for HIV-1, Vacc-4x: a phase 2 randomised, double-blind, placebo-controlled trial. Lancet Infect Dis. 2014 Apr;14(4):291-300. doi: 10.1016/S1473-3099(13)70343-8. Epub 2014 Feb 11. PMID 24525316

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was screened on 29 July 2008 and the first immunization was given on 22 August 2008. The last subject completed the study (to Week 52) on 22 June 2010. The last long-term follow-up visit was 07 June 2011.
Pre-assignment Details: 137 study participants were enrolled. One participant withdrew prior to randomization.
Groups:
- Vacc-4x Immunization (Adjuvant: GM-CSF) (Group I) While on ART: Immunization with Vacc-4x (with Leukine®) at Weeks 1, 2, 3, and 4 followed by booster immunizations at Weeks 16 and 18.
- Placebo Injections (Group II) While on ART: Placebo Vacc-4x (with placebo Leukine®) at Weeks 1, 2, 3, 4, 16 and 18.
Period: Overall Study
Arm/Group | Vacc-4x Immunization (Adjuvant: GM-CSF) (Group I) While on ART | Placebo Injections (Group II) While on ART
Started | 93 | 43
Completed | 86 | 36
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Vacc-4x Immunization (Adjuvant: GM-CSF) (Group I) While on ART | Placebo Injections (Group II) While on ART | Total
Number analyzed (Participants) | 92 | 43 | 135
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorial: <=18 years | 0 | 0 | 0
  Age, Categorial: Between 15 and 55 | 92 | 43 | 135
  Age, Categorial: >=55 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 14 | 5 | 19
  Male | 78 | 38 | 116
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 88 | 37 | 125
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height [Median (Full Range); unit: cm] | 175 [155 to 190] | 175 [159 to 200] | 175 [155 to 200]
Time since HIV diagnosis (days) [Median (Full Range); unit: days] | 3861 [466 to 8794] | 4480 [814 to 8990] | 4309 [466 to 8990]
CD4 nadir [Median (Full Range); unit: 10^6 cells/L] | 300 [200 to 734] | 285 [200 to 724] | 298 [200 to 734]
Pre-ART CD4 [Median (Full Range); unit: 10^6 cells/L] | 339 [177 to 1396] | 370 [207 to 924] | 357 [177 to 1396]
Pre-ART HIV-1 viral load [Median (Full Range); unit: copies/mL] | 94810 [120 to 2500000] | 25630 [412 to 1460000] | 75398 [120 to 2500000]
Total time on ART [Median (Full Range); unit: months] | 95.5 [13 to 276] | 112 [13 to 197] | 108 [13 to 276]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Require Resumption of ART Between the Interruption of ART at Week 28 and End of Study at Week 52.
Time Frame: From Week 28 to Week 52
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Vacc-4x Immunization (Adjuvant: GM-CSF) (Group I) While on ART | Placebo Injections (Group II) While on ART.
Number analyzed (Participants) | 92 | 43
participants
  Number of subjects attending Week 28 visit | 88 | 40
  Subjects coming off ART at Week 28 | 88 | 38
  Subjects not qualifying for ART interruption | 0 | 1
  Subjects resuming ART between week 28 and 52 | 30 | 11
  Subjects restarting ART at Week 52/termination | 12 | 7

2. Secondary Outcome: Number of Participants With Any Treatment Emergent Adverse Event, Related Treatment Emergent Adverse Events and Deaths
Description: Brief summary of treatment emergent adverse events or related treatment emergent events and deaths. The intensity of adverse events was described according to the Division of AIDS table for grading severity of adult and pediatric adverse events, 2004.
Time Frame: Up to week 52
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Vacc-4x Immunization (Adjuvant: GM-CSF) (Group I) While on ART | Placebo Injections (Group II) While on ART.
Number analyzed (Participants) | 93 | 42
participants
  Any TEAE up to week 52/early termination | 91 | 40
  TEAE - Mild | 27 | 13
  TEAE - Moderate | 54 | 21
  TEAE - Severe | 9 | 6
  TEAE - Life threatening | 1 | 0
  Related TEAE up to week 52/early termination | 81 | 24
  Related TEAE - Mild | 40 | 19
  Related TEAE - Moderate | 37 | 5
  Related TEAE - Severe | 4 | 0
  Related TEAE - Life threatening | 0 | 0
  Any TESAE up to week 52/early termination | 4 | 3
  Any related TESAE up to week 52/early termination | 1 | 0
  Any TEAE leading to treatment discontinuation | 2 | 0
  Treatment-related TEAE leading to discontinuation | 2 | 0
  Deaths | 0 | 1

3. Secondary Outcome: Immunogenicity
Description: Immunogenicity of Vacc-4x evaluated by DTH (Delayed-type Hypersensitivity) reaction. The number of participants showing induration and/or erythema
Time Frame: Week 1, week 18 and week 52
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Vacc-4x Immunization (Adjuvant: GM-CSF) (Group I) While on ART | Placebo Injections (Group II) While on ART.
Number analyzed (Participants) | 92 | 43
participants
  Induration week 1 (Vacc-4x n=92; placebo n=43 | 3 | 1
  Induration week 18 (Vacc-4x n=88; placebo n=41) | 27 | 0
  Induration week 52 (Vacc-4x n=78; placebo n=36) | 26 | 0
  Induration week 52(LOCF) Vacc-4x n=92;placebo n=43 | 30 | 0
  Erythema week 1 (Vacc-4x n=92;placebo n=43) | 3 | 1
  Erythema week 18 (Vacc-4x n=88; placebo n=41) | 40 | 0
  Erythema week 52 (Vacc-4x n=78;placebo n=36) | 34 | 0
  Erythema week 52 (LOCF) Vacc-4x n=92;placebo n=43 | 40 | 0

4. Secondary Outcome: Effect of Vacc-4x on CD8 Counts
Description: CD8 Count Over Time for subjects who stopped ART at Week 28 and remained off ART until Week 52
Time Frame: Weeks 6,18,24,28,32,36,40,44,48,52.
Population: Subject who stopped ART at week 28 and remained off ART until week 52
Measure: Median (Inter-Quartile Range); unit: cells/µL
Arm/Group | Vacc-4x Immunization (Adjuvant: GM-CSF) (Group I) While on ART | Placebo Injections (Group II) While on ART.
Number analyzed (Participants) | 56 | 25
cells/µL
  week 6 (Vacc-4x n=54;placebo n=25) | 786.0 [636.0 to 934.0] | 865.0 [544.0 to 1123.0]
  week 18 (Vacc-4x n=56; placebo n=25) | 853.5 [686.5 to 1055.0] | 897.0 [604.0 to 1176.0]
  week 24 (Vacc-4x n=56; placebo n=25) | 804.0 [583.0 to 1111.5] | 771.0 [592.0 to 1040.0]
  week 28 (Vacc-4x n=56; placebo n=25) | 820.5 [670.5 to 1050.5] | 879.0 [570.0 to 1111.0]
  week 32 (Vacc-4x n=56; placebo n=25) | 962.0 [694.5 to 1352.5] | 1161.0 [789.0 to 1456.0]
  week 36 (Vacc-4x n=56; placebo n=25) | 1385.5 [953.0 to 1748.5] | 1416.0 [1006.0 to 2058.0]
  week 40 (Vacc-4x n=54; placebo n=25) | 1252.5 [849.0 to 1788.0] | 1253.0 [866.0 to 1592.0]
  week 44 (Vacc-4x n=56; placebo n=25) | 1156.0 [799.0 to 1665.0] | 1106.0 [851.0 to 1545.0]
  week 48 (Vacc-4x n=55; placebo n=24) | 1118.0 [857.0 to 1641.0] | 1217.0 [827.0 to 1463.5]
  week 52 (completers) (Vacc-4x n=56;placebo n=25) | 1064.0 [725.0 to 1368.5] | 1047.0 [747.0 to 1502.0]

5. Secondary Outcome: Time to Restart of ART for Vacc-4x Subjects Versus Placebo
Description: Kaplan-Meier Estimate of Time to restart ART (from time coming off ART)
Time Frame: Between Week 28 to Week 52
Population: ITT Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Vacc-4x Immunization (Adjuvant: GM-CSF) (Group I) While on ART | Placebo Injections (Group II) While on ART.
Number analyzed (Participants) | 88 | 40
days | 141.8 (47.40) | 133.5 (57.27)

6. Secondary Outcome: Effects on Vacc-4x on HIV-1 RNA
Time Frame: Weeks 24,28,32,36,40,44,48,52.
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Vacc-4x Immunization (Adjuvant: GM-CSF) (Group I) While on ART | Placebo Injections (Group II) While on ART.
Number analyzed (Participants) | 92 | 43
copies/mL
  week 24 (Vacc-4x n=90; placebo n=41) | 629.6 (5807.26) | 9.2 (22.85)
  week 28 (Vacc-4x n=89; placebo n=40) | 1351.4 (5710.99) | 1628.5 (10131.81)
  week 32 (Vacc-4x n=88; placebo n=38) | 192115.0 (361003.40) | 205605.2 (383020.31)
  week 36 (Vacc-4x n=81; placebo n=35) | 89134.8 (165945.62) | 89211.9 (97983.28)
  week 40 (Vacc-4x n=71; placebo n=32) | 72705.0 (143582.93) | 76127.8 (81891.91)
  week 44 (Vacc-4x n=63; placebo n=27) | 44969.7 (65798.22) | 66203.3 (72099.23)
  week 48 (Vacc-4x n=59; placebo n=25) | 48848.2 (90232.17) | 77219.4 (70851.98)
  week 52 (Vacc-4x n=56; placebo n=24) | 35219.6 (42181.85) | 67684.0 (67869.61)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) recorded from Screening to Week 52
Description: Safety data was based on 93 Vacc-4x participants and 42 placebo participants because one placebo participant received an injection with Vacc-4x in error.
Arm/Group | Vacc-4x Immunization (Adjuvant: GM-CSF) (Group I) While on ART | Placebo Injections (Group II) While on ART
Serious Adverse Events (participants affected / at risk) | 4/93 | 3/42
Other Adverse Events (participants affected / at risk) | 91/93 | 40/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vacc-4x Immunization (Adjuvant: GM-CSF) (Group I) While on ART (N=93) | Placebo Injections (Group II) While on ART (N=42)
Appendicitis perforated (Gastrointestinal disorders) | 1 (1) | 0 (0) — Perforated appendix
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0) — Multiple sclerosis
Cellulitis of male external genital organ (Infections and infestations) | 1 (1) | 0 (0) — Cellulitis of scrotum and penis
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) — Acute appendicitis resulting in appendectomy
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) — Surgical wound infection
Necrosis (General disorders) | 0 (0) | 1 (1) — Atypic(al) necrosis of both femoral heads
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1) — Bipolar disorder resulting in hospitalization
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Prolonged anesthesia effects (dizziness)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vacc-4x Immunization (Adjuvant: GM-CSF) (Group I) While on ART (N=93) | Placebo Injections (Group II) While on ART (N=42)
Injection site erythema (General disorders) | 62 | 6 — Injection site erythema
Injection site induration (General disorders) | 39 | 6
Injection site pruritus (General disorders) | 35 | 0
Fatigue (General disorders) | 11 | 5
Injection site pain (General disorders) | 16 | 6
Pyrexia (General disorders) | 7 | 1
Injection site swelling (General disorders) | 15 | 3
Nasopharyngitis (Infections and infestations) | 5 | 0
Nausea (Gastrointestinal disorders) | 4 | 2
Headache (Nervous system disorders) | 7 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 1
Influenza-like illness (General disorders) | 3 | 1
Asthenia (General disorders) | 4 | 0
Chills (General disorders) | 4 | 0
Malaise (General disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 1
ALT increased (Investigations) | 0 | 1
AST increased (Investigations) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor (or designee) will prepare a final report on the study. The Investigator may not publish or present any information on this study without the express written approval of the Sponsor. Additionally, the Sponsor, may, for any reason, withhold approval for publication or presentation.